CLINICAL TRIAL: NCT00888667
Title: Optimal EGM Configuration for Morphology Discrimination
Acronym: SVT Morphology
Status: Terminated | Type: Observational
Why Stopped: Patient population was not available
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: HV001
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Premature Ventricular Complexes
Keywords: ICD patients with PVCs and EGM recordings
MeSH Terms: conditions — Ventricular Premature Complexes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICD patient with frequent PVCs
  Interventions: Other: Pacing interventions

INTERVENTIONS:
Other: Pacing interventions — 10 seconds recording of atrial paced rhythm at 100 ppm in sitting 10 seconds recording of atrial paced rhythm at 150 ppm in supine 10 seconds recording of atrial paced rhythm at 150 ppm in sitting

SUMMARY:
The study will be a prospective cohort study of 20 patients recruited from site's Defibrillator Clinic patient population who are followed at the site.

Hypothesis: Among the available EGM configuration options, one is better than the others for detection enhancements purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must already have an implanted St. Jude Medical dual chamber ICD with a dual coil defibrillator lead.
2. Patients must be willing to sign an informed consent form.
3. Patients must have frequent PVCs (minimum of 30/hour)

Exclusion Criteria:

1. Known history of slow VT (under 160 bpm).
2. Patients under the age of 18 years.
3. Pregnant women.
4. Pacemaker dependent rhythm.
5. Ongoing angina pectoris.
6. Current NYHA Class 3-4 heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a dual chamber ICD and frequent PVCs
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
% morphology match | acute
  off line analysis

CONTACTS AND LOCATIONS:
Locations (1):
- St Michael's Hospital, Toronto, Ontario, Canada